CLINICAL TRIAL: NCT06938243
Title: The Comparison of Safety and Treatment Results Between Early (<6 Months) and Late (> 6 Months) Vagus Stimulation for Post-stroke Motor Rehabilitation: a Randomized Clinical Trial
Brief Title: Wether VNS in Early Stage (3 Months) is Safe and More Beneficial for Post-stroke Motor Rehabilitation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Early VNS for Motor Rehabilita
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Motor Rehabilitation
Keywords: Hemiparesis; VNS; Limb Motor Function Rehabilitation
MeSH Terms: conditions — Stroke; Paresis | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- VNS activated in late stage (Experimental): Following enrollment, participants with a history of stroke greater than 6 months underwent 1 month of upper-extremity rehabilitation twice per week to rule out potential for recovery with rehabilitation therapy alone. Thereafter, each participant underwent surgical implantation of the VNS system. 1 months later, VNS was activated.
  Interventions: Device: Vagus Nerve Stimulation in late stage
- VNS activated in early stage (Active Comparator): Following enrollment, participants with a history of stroke within 6 months underwent 1 month of upper-extremity rehabilitation twice per week to rule out potential for recovery with rehabilitation therapy alone. Thereafter, each participant underwent surgical implantation of the VNS system. 1 months later, VNS was activated.
  Interventions: Device: Vagus Nerve Stimulation in early stage
- VNS not activated in early stage (Experimental): Following enrollment, participants with a history of stroke within 6 months underwent 1 month of upper-extremity rehabilitation twice per week to rule out potential for recovery with rehabilitation therapy alone. Thereafter, each participant underwent surgical implantation of the VNS system.When the a history of stroke was exceeded over 6 months, VNS was activated.
  Interventions: Device: Vagus Nerve Stimulation in late stage

INTERVENTIONS:
Device: Vagus Nerve Stimulation in early stage — Device implantation was done under general anaesthesia. A horizontal neck crease incision was created left of the midline at the level of the cricoid cartilage. After the vagus nerve was identified, the stimulation lead was wrapped around the vagus nerve. The lead was then tunnelled subcutaneously to the pulse generator device which was contained in a subcutaneous pocket in the pectoral region.
  Arms: VNS activated in early stage
Device: Vagus Nerve Stimulation in late stage — Device implantation was done under general anaesthesia. A horizontal neck crease incision was created left of the midline at the level of the cricoid cartilage. After the vagus nerve was identified, the stimulation lead was wrapped around the vagus nerve. The lead was then tunnelled subcutaneously to the pulse generator device which was contained in a subcutaneous pocket in the pectoral region
  Arms: VNS activated in late stage; VNS not activated in early stage

SUMMARY:
Upper-extremity impairment after stroke remains a major therapeutic challenge and a target of neuromodulation treatment efforts. In previous study, Vagus nerve stimulation was constricted to patients 9 months after stroke. In this randomized phase I trial, we would apply vagus nerve stimulation in an early stage (<6 month) and observe its theraputic effect on motor function after ischaemic Stroke.We hypothesized that the early stimulation could be safe and more beneficial compared to stimulation in late stage.

ELIGIBILITY:
Inclusion Criteria:

* Eligible individuals suffered a first-time, unilateral, ischemic stroke in the middle cerebral artery territory that spared the diencephalon and basal ganglia 3-36 months before surgery.

  * Individuals with persistent moderate-to-severe upper-extremity hemiparesis as defined by an FM-UE score of ≤42
  * Sufficient upper-extremity motor ability to engage in rehabilitation (that is, a score of ≥1 on the FM-UE elbow flexion, elbow extension or finger mass flexion or extension).

Exclusion Criteria:

* Excessive spasticity or contracture of the upper-extremity muscles (that is, Modified Ashworth Scale = 4) . Severe cognitive impairment (Mini Mental State Examination < 24)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
FM-UE scores between early and late VNS | 12 months after device implantation
  The outcomes includes each participant's Fugl-Meyer assessment scale (FM-UE) scores for each monthly visit. FM-UE scores range from 0 to 100 and the higher scores indicated better outcome of movement.

SECONDARY OUTCOMES:
Arm Motor Ability Test (AMAT) between early and late VNS | 12 months after device implantation
  The outcomes includes each participant's the Arm Motor Ability Test (AMAT) for each monthly visit. AMAT scores range from 0 to 57 and the higher scores indicated better outcome of movement.
the Nine-Hole Peg Test between early and late VNS | 12 months after device implantation
  The outcomes includes each participant's the Nine-Hole Peg Test for each monthly visit.
the Bilateral Box and Block Test between early and late VNS | 12 months after device implantation
  The outcomes includes each participant's the Bilateral Box and Block Test for each monthly visit.
Short Form Health Survey (SF-12) between early and late VNS | 12 months after device implantation
  The outcomes includes each participant's score of Short Form Health Survey (SF-12) for each monthly visit. SF-12 scores range from 0 to 60 and the higher scores indicated better outcome of movement.
the EuroQol Five Dimensions Questionnaire (EQ-5D) between early and late VNS | 12 months after device implantation
  The outcomes includes each participant's score of the EuroQol (EQ-5D) scores range from 0 to 36 for each monthly visit.
safety and feasibility of early and late VNS | 12 months after device implantation
  The incidence of adverse events including hemorrhages, infections, deaths or major perioperative complications during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP